CLINICAL TRIAL: NCT01620177
Title: Effects of Inhaled Cannabis on Driving Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary R Gaffney (Other)
Collaborators: National Highway Traffic Safety Administration (NHTSA) (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Gary R Gaffney, Associate Professor, College of Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 201109850
Record Dates: First submitted 2012-06-04; First posted 2012-06-15 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Alcohol Drinking; Cannabis
Keywords: Cannabis; Marijuana; Marihuana; Alcohol; Driving
MeSH Terms: conditions — Alcohol Drinking; Marijuana Abuse | interventions — Ethanol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 0% THC with 0.065 g/dL BAC (Experimental)
  Interventions: Drug: Alcohol(oral) and placebo; Drug: Cannabis(THC)(Inhaled) and Placebo
- 2.5-3.5% THC with 0.065 g/dL BAC (Experimental)
  Interventions: Drug: Alcohol(oral) and placebo; Drug: Cannabis(THC)(Inhaled) and Placebo
- 6.0-7.5% THC and 0.065 g/dL BAC (Experimental)
  Interventions: Drug: Alcohol(oral) and placebo; Drug: Cannabis(THC)(Inhaled) and Placebo
- 2.5-3.5% THC with 0 g/dL BAC (Experimental)
  Interventions: Drug: Alcohol(oral) and placebo; Drug: Cannabis(THC)(Inhaled) and Placebo
- 6.0-7.5% THC with 0 g/dL BAC (Experimental)
  Interventions: Drug: Alcohol(oral) and placebo; Drug: Cannabis(THC)(Inhaled) and Placebo
- 0% THC with 0 g/dL BAC (Experimental)
  Interventions: Drug: Alcohol(oral) and placebo; Drug: Cannabis(THC)(Inhaled) and Placebo

INTERVENTIONS:
Drug: Alcohol(oral) and placebo — Subjects will be dosed to an approximate peak BAC of 0.065%. Subjects will be tested on the decline such that subjects will be at or above the goal BAC (0.05%) throughout the drive
  Other Names: Ethanol; Ethyl Alcohol
Drug: Cannabis(THC)(Inhaled) and Placebo — Cannabis vapor is produced from 500 mg either placebo (0% THC), approximately 2.5-3.5% THC (low dose), or approximately 6.0-7.5% THC (high dose) bulk cannabis plant material to yield doses of approximately 0, 12.5-17.5, or 30-37.5 mg THC
  Other Names: Marihuana; Marijuana

SUMMARY:
The purpose of this study is to expand understanding of the effects of cannabis on driving performance with and without the presence of low levels of alcohol.

This project will involve the development a of a protocol and driving environment that is sensitive to the effects of cannabis on driving performance by building on prior driving situations used previously for testing the effects of alcohol on driving.

DETAILED DESCRIPTION:
Individuals will be recruited who are currently users of cannabis and alcohol to participate in this study. They will undergo a physical exam at screening. There will be six study visits where the subject will arrive at the Clinical Research Unit(University of Iowa Hospitals & Clinics) the night before dosing. At each visit subjects will be receive one of the following six dosing regimens: placebo alcohol with placebo cannabis; placebo alcohol with low-dose cannabis, placebo alcohol with higher-dose of cannabis, low dose alcohol with placebo cannabis; low dose alcohol with low dose cannabis, low dose alcohol with higher-dose of cannabis. After dosing, participants will have provide saliva samples and blood drawn periodically to check cannabis levels and will complete a driving simulation. After completing the drive, additional saliva samples and blood draws will occur and participants will be monitored until it is safe to transport home.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult (age 21-55) men and women, based on medical and psychological evaluation
* Currently valid unrestricted (except for vision correction) US driver's license
* Licensed driver for at least the past two years
* Drove at least 1300 miles in the past year, by self-report
* Live within an 80 mile radius of NADS
* Available for an overnight stay followed by a full-day study session for six sessions
* Must be considered a light or moderate drinker according to Quantity-Frequency-Variability Scale (QFV)
* Cannabis use with a minimum frequency averaging at least one day per quarter and no more than three days a week during the three months prior to study entry
* Peripheral veins suitable for repeated venipuncture and/or placement of an intravenous catheter
* Systolic blood pressure within a clinically normal range (120 ± 30 mmHg) and -diastolic blood pressure of 80 ± 20 mmHg..
* Good command of written and spoken English
* Female subjects with reproductive potential must agree to use (and/or have their partner use) one (1) acceptable method of birth control beginning at the screening visit throughout the study (including intervals between treatment periods/panels) and until 2 weeks after the last dose of study drug in the last treatment period. Acceptable methods of birth control include the following: intrauterine device (IUD-with or without local hormone release), diaphragm, spermicides, cervical cap, contraceptive sponge, oral contraceptives or condoms. Abstinence is an alternative lifestyle and subjects practicing abstinence may be included in the study.

Exclusion Criteria:

* Presence of any clinically significant illness, as detected by history, physical examination, and/or laboratory tests, that might influence driving performance (e.g., seizures, sleep apnea, narcolepsy, vertigo, chronic fatigue syndrome) or put the subject at increased risk of adverse events (e.g., cardiac arrhythmia, hypertension)
* History of a clinically significant adverse event associated with cannabis or alcohol intoxication
* Donation of more than 450 mL of blood within 14 days of study drug administration
* If female, pregnant or nursing
* Currently interested in or participating in drug abuse treatment, or participated in drug abuse treatment within 60 days preceding study enrollment
* Currently taking drugs that are contraindicated for use with study drugs
* Requires any special equipment to aid in driving (ex. pedal extensions, hand brake or throttle, spinner wheel knobs or other non-standard equipment)
* Significant history of motion sickness or demonstrates significant simulator sickness during practice drives at screening (SSQ). Subjects must have scores below the following values on the SSQ: Nausea < 21, Oculomotor <32, Disorientation < 15, and Total Score < 32.
* Current alcohol or cannabis use disorder, as identified by the Alcohol Use Disorders Identification Test for alcohol or Cannabis Use Disorders Identification Test for cannabis.
* History of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the subject from study participation
* Prior participation in a driver impairment or distraction-related research study conducted at NADS that uses the same base drive.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary G Gaffney, M.D., Principal Investigator — National Advanced Driving Simulator
Locations (1):
- National Advanced Driving Simulator, Iowa City, Iowa, United States

REFERENCES:
- [Result] Hartman RL, Brown TL, Milavetz G, Spurgin A, Pierce RS, Gorelick DA, Gaffney G, Huestis MA. Cannabis effects on driving lateral control with and without alcohol. Drug Alcohol Depend. 2015 Sep 1;154:25-37. doi: 10.1016/j.drugalcdep.2015.06.015. Epub 2015 Jun 23. PMID 26144593
- [Result] Hartman RL, Brown TL, Milavetz G, Spurgin A, Gorelick DA, Gaffney G, Huestis MA. Controlled Cannabis Vaporizer Administration: Blood and Plasma Cannabinoids with and without Alcohol. Clin Chem. 2015 Jun;61(6):850-69. doi: 10.1373/clinchem.2015.238287. Epub 2015 May 27. PMID 26019183
- [Result] Hartman RL, Brown TL, Milavetz G, Spurgin A, Gorelick DA, Gaffney G, Huestis MA. Controlled vaporized cannabis, with and without alcohol: subjective effects and oral fluid-blood cannabinoid relationships. Drug Test Anal. 2016 Jul;8(7):690-701. doi: 10.1002/dta.1839. Epub 2015 Aug 10. PMID 26257143
- [Result] Hartman RL, Brown TL, Milavetz G, Spurgin A, Pierce RS, Gorelick DA, Gaffney G, Huestis MA. Cannabis effects on driving longitudinal control with and without alcohol. J Appl Toxicol. 2016 Nov;36(11):1418-29. doi: 10.1002/jat.3295. Epub 2016 Feb 18. PMID 26889769

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Individuals who completed the study completed all six arms of the study and the data is aggregated. Non-completers may have completed some arms and not others and their data is aggregated. There will be six study visits where the subject will arrive at the Clinical Research Unit(University of Iowa Hospitals & Clinics) the night before dosing. At each visit subjects will be receive one of the following six dosing regimens: placebo alcohol with placebo cannabis; placebo alcohol with low-dose cannabis, placebo alcohol with higher-dose of cannabis, low dose alcohol with placebo cannabis; low dose alcohol with low dose cannabis, low dose alcohol with higher-dose of cannabis.
Period: Overall Study
Arm/Group | Overall Study
Started | 98
Completed | 19
Not Completed | 79
Not completed — Failure at Screening Visit | 43
Not completed — Withdrawal by Subject | 26
Not completed — Lost to Follow-up | 7
Not completed — Physician Decision | 2
Not completed — Randomized, Not Active due to Scheduling | 1

BASELINE CHARACTERISTICS:
Population: There was no baseline group, but rather all subjects who completed experienced the baseline dosing condition of placebo cannabis and placebo alcohol.
Groups:
- Overall Study: Individuals who completed the study completed all six arms of the study and the data is aggregated. Non-completers may have completed some arms and not others and their data is aggregated.
Arm/Group | Overall Study
Number analyzed (Participants) | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 98
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 89
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 84
  More than one race | 6
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 98

OUTCOME MEASURES:

1. Primary Outcome: Driving Performance
Description: Measured by standard deviation of lane position. Metrics of driving performance were modeled using the SAS GLM Select function to identify changes in driver performance. Numbers represents coefficients on the regression equation such that this increase would be expected for every unit increase. A unit for THC is 1 ng/ml and a unit for BAC is 0.01% BAC. In understanding the regression coefficients, for THC the units for the coefficient would be expressed as cm per (ng/ml of THC), and for BrAC the units for the coefficient would be expressed as cm per (0.01% BrAC). The overall regression equation would be represented as SDLP = Intercept + Cthc x THC + Cbrac x BrAC. The coefficients indicate the strength of the effect on driving performance with higher coefficients indicating larger effects relative to the concentrations. Coefficients of zero indicate no effect or interactive effect.
Time Frame: Through entire drive, 0.5-1.3 hr post cannabis administration.
Population: One subject who was an extreme outlier across driving performance measures was excluded. Due to the variability in THC and BrAC levels across subjects and conditions, a regression model was used which combined all of the data.
Measure: Number; unit: cm
Groups:
- Cannabis - THC: Data from all dosing conditions combined to estimate the effect of THC concentrations using a regression equation.
- Alcohol - BrAC (Breath Alcohol Concentration): Data from all dosing conditions combined to estimate the effect of BrACconcentrations using a regression equation.
- THC x BrAC: Data from all dosing conditions combined to estimate the interactive effect of THC and BrAC concentrations using a regression equation.
Arm/Group | Cannabis - THC | Alcohol - BrAC (Breath Alcohol Concentration) | THC x BrAC
Number analyzed (Participants) | 18 | 18 | 18
cm | 0.26 | 0.42 | 0

2. Secondary Outcome: THC Concentration in Plasma Sample
Description: Measurement of THC concentration levels in plasma over the course of each visit compared to that of the other visits.
Time Frame: -0.7 hr, 0.25hr, 1.1 hr, 2 hr, 3 hr, 4.5 hr, 6 hr, 8 hr post cannabis administration
Population: We performed noncompartmental analyses with Phoenix WinNonLin® 6.3 for Windows (Pharsight) for maximum concentration (Cmax) of 11-OH-THC (LOQ 1 μg/L).
Measure: Median (Full Range); unit: ng/ml
Arm/Group | 0% THC With 0.065 g/dL BAC | 2.5-3.5% THC With 0.065 g/dL BAC | 6.0-7.5% THC and 0.065 g/dL BAC | 2.5-3.5% THC With 0 g/dL BAC | 6.0-7.5% THC With 0 g/dL BAC | 0% THC With 0 g/dL BAC
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
ng/ml | 0 [0 to 3.2] | 4.8 [1.3 to 8] | 7.5 [0 to 27.3] | 4.1 [0 to 13.7] | 7 [1.0 to 20.3] | 0 [0 to 4.3]

3. Secondary Outcome: THC Concentration Levels in Whole Blood
Description: Measurement of THC concentration levels in whole blood over the course of each visit compared to that of the other visits.
Time Frame: -0.7 hr, 0.25hr, 1.1 hr, 2 hr, 3 hr, 4.5 hr, 6 hr, 8 hr post cannabis
Measure: Median (Full Range); unit: ng/ml
Arm/Group | 0% THC With 0.065 g/dL BAC | 2.5-3.5% THC With 0.065 g/dL BAC | 6.0-7.5% THC and 0.065 g/dL BAC | 2.5-3.5% THC With 0 g/dL BAC | 6.0-7.5% THC With 0 g/dL BAC | 0% THC With 0 g/dL BAC
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
ng/ml | 0 [0 to 2.4] | 3.7 [1.4 to 6.0] | 6.0 [0 to 24.8] | 2.8 [0 to 9.1] | 5.0 [0 to 14.2] | 0 [0 to 2.5]

ADVERSE EVENTS:
Description: Adverse events were reported for all subjects who completed at least one dosing visit. The number of subjects varies across conditions based on the number of dosing visits by subjects who did not complete the study and which randomization arm they were assigned.
Arm/Group | 0% THC With 0.065 g/dL BAC | 2.5-3.5% THC With 0.065 g/dL BAC | 6.0-7.5% THC and 0.065 g/dL BAC | 2.5-3.5% THC With 0 g/dL BAC | 6.0-7.5% THC With 0 g/dL BAC | 0% THC With 0 g/dL BAC
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27 | 0/24 | 0/26 | 0/31 | 0/27
Other Adverse Events (participants affected / at risk) | 4/29 | 4/27 | 6/24 | 0/26 | 3/31 | 0/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0% THC With 0.065 g/dL BAC (N=29) | 2.5-3.5% THC With 0.065 g/dL BAC (N=27) | 6.0-7.5% THC and 0.065 g/dL BAC (N=24) | 2.5-3.5% THC With 0 g/dL BAC (N=26) | 6.0-7.5% THC With 0 g/dL BAC (N=31) | 0% THC With 0 g/dL BAC (N=27)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tooth Ache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — This AE was the result of wisdom teeth pain, and the participant subsequently had the teeth removed.
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of Consciousness with IV Insertion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Light-Headed (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change in Status Perception (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diaphoresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study examined only occasional users and the generalization to new or frequent cannabis users is unclear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days